CLINICAL TRIAL: NCT00561379
Title: Frontline Therapy of Diffuse Large B Cell Lymphoma of the Adult ( 18 to 60 Years Old): Randomization Between High Dose Chemotherapy With Rituximab and CHOP 14 -Rituximab. Multicentric Randomized Prospective Trial.
Brief Title: Diffuse Large B Cell Lymphoma of the Adult: Randomization Between High Dose Chemotherapy With Rituximab and CHOP 14-Rituximab
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BRD 04/4-O
Record Dates: First submitted 2007-11-20; First posted 2007-11-21 (Estimated); Last update posted 2013-06-13 (Estimated); Status verified 2013-06

CONDITIONS: Lymphoma, Large-Cell, Diffuse
Keywords: Diffuse Large B Cell Lymphoma; not previously treated
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse

ARMS (2):
- 1 (Active Comparator)
  Interventions: Drug: CHOP+RITUXIMAB
- 2 (Active Comparator)
  Interventions: Drug: CEEP-RITUXIMAB

INTERVENTIONS:
Drug: CHOP+RITUXIMAB — CHOP-14- Rituximab x 8 courses
  Arms: 1
Drug: CEEP-RITUXIMAB — High dose chemotherapy with rituximab including autologous stem cell support.
  Arms: 2

SUMMARY:
The aim of the protocol is to compare the outcome of patients with DLBCL stage II bulky, III or IV with 1 to 3 adverse prognostic factors according to the International prognostic index. Patients with eligibility criteria and who gave informed consent will be randomised between CHOP-14- Rituximab x 8 courses and High dose chemotherapy with rituximab including autologous stem cell support. The aim of the study is to compare the Event free survival between the two arms and to gain insight into the prognostic significance of several biological markers gathered at the time of diagnosis/randomisation ( i.e. Fcgamma R III A genotyping, DNA profile and BCL é expression).

DETAILED DESCRIPTION:
Diffuse Large B Cell Lymphoma not previously treated

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 et ≤ 60 and male and female
* Diffuse large B cell lymphoma according to WHO classification phénotype B CD 20 +
* Stage I et II tumor bulk > 7 cm and stage III et IV Ann Arbor.
* Non previously treated
* HIV négative
* Signed informed consent

Exclusion Criteria:

* Age < 18 and/or > 60 ans
* NHL not DLBCL
* Lymphoblastic Lymphoma
* Burkitt's Lymphoma
* Low grade Lymphoma transformed
* Primary CNS Lymphomal
* Post- transplantation Lymphoma
* CD20 negative
* Ann Arbor stage I or II without tumor bulk > 7 cm
* Previous treatment
* HIV positive
* Contre-indication to Rituximab use according to SmPC
* Contre-indication to high dose chemotherapy due to organ failure not related to the lymphoma
* Cancer or history of cancer with the exception of in situ cancer of the cervix or non-invasive skin epithelioma
* Patient not able to understand the proposed treatments
* Refusal to sign the informed consent

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 350 (Estimated)
Dates: Start 2005-04; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
3 years Event-free survival ( Kaplan Meier method)

SECONDARY OUTCOMES:
3 years overall survival
Prognostic impact of: Level of expression of protéine bcl2 protein in tumor cells; FCGR3A genotype; génomic profile (DNA microarray)on response, survival, and Event-Free-Survival
Cost

CONTACTS AND LOCATIONS:
Overall Officials: Noel Milpied, MD, Principal Investigator — University Hospital, Bordeaux
Locations (1):
- Nantes University Hospital, Nantes, France